CLINICAL TRIAL: NCT02722837
Title: A Phase 3, Open-label Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Subjects With Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination in Participants With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1522; 2015-003001-42 (EudraCT Number)
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SOF/VEL (Experimental): SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®

SUMMARY:
The primary objective of this study is to evaluate the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) for 12 weeks in participants with chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* HCV RNA ≥ 10^4 IU/mL at screening
* Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy

Key Exclusion Criteria:

* Any other chronic liver disease
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Clinical hepatic decompensation
* Prior exposure to SOF or other nucleotide analogue HCV NS5B inhibitor or any HCV NS5A inhibitor

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (15):
- Russia (13):
  - Krasnoyarsk Regional Center of AIDS Prevention, Krasnoyarsk
  - Central Research Institute of Epidemiology, Moscow
  - Central Scientific-Research Institute of Epidemiology, Moscow
  - City Clinical Hospital # 24, Moscow
  - First Moscow Medical University I.M.Sechenov., Moscow
  - First Moscow State Medical University I.M. Sechenov, Moscow
  - Limited Liability Company "Clinic Tour", Moscow
  - Scientific Research Institute of Nutrition, Moscow
  - Sklifosovsky Scientific Research Institution of Emergency Care, Moscow
  - Center for Prevention and Control of AIDS and Infectious Diseases, Saint Petersburg
  - Kirov Medical Military Academy, Saint Petersburg
  - North-Western State Medical University named after I.I. Mechnikov, Saint Petersburg
  - LLC Medical Company "Hepatolog", Samara
- Sweden (2):
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Karolinska University Hospital Huddinge, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Background] Weiland O, Zhdanov K, Chulanov VP, McNabb BL, Lu S, Svarovskaia EU, et al. Safety and Efficacy of Sofosbuvir/Velpatasvir in a Genotype 1-3 HCV Infected Russian and Swedish Population: Results from a Phase 3, Prospective Trial [Abstract 1186]. Hepatology 2017;66 (1):639A.
- [Derived] Isakov V, Chulanov V, Abdurakhmanov D, Burnevich E, Nurmukhametova E, Kozhevnikova G, Gankina N, Zhuravel S, Romanova S, Hyland RH, Lu S, Svarovskaia ES, McNally J, Brainard DM, Ivashkin V, Morozov V, Bakulin I, Lagging M, Zhdanov K, Weiland O. Sofosbuvir/velpatasvir for the treatment of HCV: excellent results from a phase-3, open-label study in Russia and Sweden. Infect Dis (Lond). 2019 Feb;51(2):131-139. doi: 10.1080/23744235.2018.1535186. Epub 2018 Nov 30. PMID 30499360

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the Russian Federation and Sweden. The first participant was screened on 04 April 2016 and the last study visit occurred on 13 September 2017.
Pre-assignment Details: 122 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet administered orally once daily for 12 weeks, with or without food
Period: Overall Study
Arm/Group | SOF/VEL
Started | 119
Completed | 119
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet administered orally once daily for 12 weeks, with or without food
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  White | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 119
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 16
  Russia | 103
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 29
    CT | 72
    TT | 18
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.1 (0.54)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 38
  ≥ 800,000 IU/mL | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 99.2 [95.4 to 100.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 100.0 [96.6 to 100.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 99.2 [95.4 to 100.0]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment at Week 1
Time Frame: Week 1
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 21.0 [14.1 to 29.4]

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment at Week 2
Time Frame: Week 2
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 64.7 [55.4 to 73.2]

7. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment at Week 4
Time Frame: Week 4
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 96.6 [91.6 to 99.1]

8. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment at Week 8
Time Frame: Week 8
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 100.0 [96.9 to 100.0]

9. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment at Week 12
Time Frame: Week 12
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 100.0 [96.9 to 100.0]

10. Secondary Outcome: Change From Baseline in HCV RNA at Week 1
Time Frame: Baseline (Day 1); Week 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 118
log10 IU/mL | -4.17 (0.502)

11. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline (Day 1); Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 117
log10 IU/mL | -4.70 (0.525)

12. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline (Day 1); Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
log10 IU/mL | -4.90 (0.540)

13. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline (Day 1); Week 8
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
log10 IU/mL | -4.93 (0.544)

14. Secondary Outcome: Change From Baseline in HCV RNA at Week 12
Time Frame: Baseline (Day 1); Week 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
log10 IU/mL | -4.93 (0.544)

15. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment), or
  * Relapse (HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement)
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 119
percentage of participants | 0.8

ADVERSE EVENTS:
Time Frame: Up to 12 weeks + 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL
All-Cause Mortality (participants affected / at risk) | 0/119
Serious Adverse Events (participants affected / at risk) | 4/119
Other Adverse Events (participants affected / at risk) | 29/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=119)
Orchitis (Infections and infestations) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Sciatica (Nervous system disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=119)
Asthenia (General disorders) | 7
Fatigue (General disorders) | 8
Headache (Nervous system disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02722837/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT02722837/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02722837/SAP_002.pdf